CLINICAL TRIAL: NCT06801405
Title: Antibiotic Prophylaxis in Percutaneous Nephrostomy Placements and Replacements for Malignant Urinary Tract Obstruction. A Retrospective Cohort Study
Brief Title: Antibiotic Prophylaxis in Percutaneous Nephrostomy Placements and Replacements for Malignant Urinary Tract Obstruction
Status: Completed | Type: Observational
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Principal Investigator, Jeferson Rodrigo Zanon, Principal Investigator, Barretos Cancer Hospital
Other Study IDs: 44395921.4.0000.5437
Record Dates: First submitted 2025-01-18; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Ureteral Obstruction; Neoplasms; Acute Kidney Injury; Nephrostomy; Complications; Antibiotic Prophylaxis; Urinary Tract Infections
Keywords: antibiotic prophylaxis; percutaneous nephrostomy; urinary tract infections; cancer patients
MeSH Terms: conditions — Ureteral Obstruction; Neoplasms; Acute Kidney Injury; Urinary Tract Infections | interventions — Antibiotic Prophylaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- No antibiotic prophylaxis (NAP) - Group: No antibiotic prophylaxis before percutaneous nephrostomy
- Antibiotic prophylaxis (AP) - Group: With antibiotic prophylaxis before percutaneous nephrostomy
  Interventions: Drug: antibiotic prophylaxis

INTERVENTIONS:
Drug: antibiotic prophylaxis — Antibiotic prophylaxis before percutaneous nephrostomy
  Groups: Antibiotic prophylaxis (AP) - Group

SUMMARY:
This study aims to find out whether taking antibiotics to prevent a urinary tract infection after a medical procedure called percutaneous nephrostomy (placement of a catheter directly into the kidney to keep it working after the urinary tract has been blocked by a malignant tumour) actually prevents a urinary tract infection, compared to not taking antibiotic prophylaxis.

DETAILED DESCRIPTION:
The medical records of cancer patients who underwent percutaneous nephrostomy between January 2013 and July 2020 were reviewed. Procedures were excluded if the nephrostomy was used for other procedures (e.g. double-J passage) or for non-malignant urinary tract obstruction (e.g. kidney stones). The association between antibiotic prophylaxis and UTI was assessed using association tests such as Pearson's chi-squared or Fisher's exact test. A significant level of 5% was adopted.

Definitions:

Urinary tract infection - occurs when there are signs and symptoms consistent with a local infection (fever, chills, dysuria, lower back pain, and costovertebral angle tenderness), such as cystitis (bladder or lower UTI) or pyelonephritis (kidney or upper UTI), combined with a positive urine culture (more than 104 colony-forming units of microorganisms per millilitre of urine with a catheter present or more than 105 colony-forming units of microorganisms per millilitre of urine without a catheter present).

UTI related to percutaneous nephrostomy procedure - occurs until seven days after the percutaneous nephrostomy procedure, both for first placement and/or catheter replacement.

UTI related to the nephrostomy catheter - occurs at another time, usually within 90 days of the procedure, in the presence of the nephrostomy catheter, and in the absence of another focus that would justify the infection.

Antibiotic prophylaxis was administered before percutaneous nephrostomy. If there was no record of antibiotics in the cost centre of the institution's database, it was considered that antibiotic prophylaxis was not given.

For the first percutaneous nephrostomy catheter placement, antibiotic prophylaxis was given empirically.

For catheter replacement, antibiotic prophylaxis was both empirical and targeted, based on the result of a pre-procedure urine culture to guide the antibiotic choice.

Percutaneous nephrostomies (first placement and/or catheter replacement) were excluded from analysis if patients were treated for UTI up to 7 days before or during the procedure. However, they were included in analysis outside the period of antibiotic prophylaxis for future UTIs.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for cancer who required percutaneous nephrostomies

Exclusion Criteria:

* Patients and/or procedures if percutaneous nephrostomy was used to perform other procedures;
* Patients and/or procedures if percutaneous nephrostomy was used to treat clinical conditions other than malignant ureteral obstruction
* Patients and/or procedures if percutaneous nephrostomy was used to clear the urinary tract of non-malignant causes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated for cancer who required percutaneous nephrostomies
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2021-04-02 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Urinary tract infection rate | Up to 7 days after percutaneous nephrostomy
  Proportion of urinary tract infection after each percutaneous nephrostomy

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo RD Reis, Study Chair — Barretos Cancer Hospital
Locations (1):
- Jales Cancer Hospital, Jales, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Publication in a peer-reviewed journal and release of data upon plausible justification
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: For an indefinite period
Access Criteria: Justification sent by e-mail